CLINICAL TRIAL: NCT06715332
Title: Safety and Efficacy of the Novel SpydrBlade Flex With Radiofrequency and Microwave Ablation Flexible Bipolar for Colorectal Endoscopic Submucosal Dissection - A Prospective Study
Brief Title: Prospective Study of Using Novel Bipolar Scissors in Colorectal Endoscopic Submucosal Dissection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2024.495
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Colon Polyp; Colon Neoplasia
Keywords: Endoscopic submucosal dissection
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic submucosal dissection with SpydrBlade Flex (Experimental): This group of patient would undergo endoscopic submucosal dissection with the use of the novel SpydrBlade Flex knife
  Interventions: Device: Colorectal ESD with SpydrBlade Flex

INTERVENTIONS:
Device: Colorectal ESD with SpydrBlade Flex — The allocated intervention would be performed under sedation or monitored anaesthesia by experienced endoscopists with at least 50 case experience of colon ESD.
  Colon ESD procedure would be performed as per described in the literature. After submucosal injection of solution to create a cushion, mucosal incision and submucosal dissection would be performed with the SydrBlade Flex. Submucosal plane dissection will be performed using the SpydrBlade Flex (BRF, cutting frequency 400kHz, power setting 35W). The exact resection strategy would be according to the endoscopists' preference, including different adjunctive techniques such as countertraction, tunnelling or pocket creation method. Upon completion of ESD, the resultant mucosal defect would be examined for any perforation or bleeding.

SUMMARY:
This study is an interventional, prospective, single-center study to evaluate the safety and effectiveness of a novel radiofrequency and microwave ablation flexible bipolar (SpydrBlade Flex, CREO Medical, UK) for colorectal ESD in patients with superficial colorectal neoplasia.

DETAILED DESCRIPTION:
This is a prospective study with the following study Objectives:

1. To evaluate the safety and effectiveness of a novel radiofrequency and microwave ablation flexible bipolar (SpydrBlade Flex, CREO Medical, UK) for colorectal ESD.
2. To assess the impact of the procedure on patient recovery time and postoperative adverse event.

This study is an interventional, prospective, single-center study to evaluate the safety and effectiveness of a novel radiofrequency and microwave ablation flexible bipolar (SpydrBlade Flex, CREO Medical, UK) for colorectal ESD in patients with superficial colorectal neoplasia. Patients will undergo a ESD for superficial colorectal neoplasia. All ESD procedures will be performed by expert endoscopists with at least 50 prior experience of ESD.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (age ≥18 and ≤80 years-old)
* Capability of understanding and complying with the study requirements, including signing the informed consent form.
* Patients with colorectal superficial mucosal neoplasia (clinically adenoma or early intramucosal cancer), scheduled to undergo endoscopic submucosal dissection (ESD).

Exclusion criteria:

* Patients unable or unwilling to provide consent.
* Patients with lesions unsuitable for ESD, including those suspicious of deep submucosal invasive cancer.
* Patients with lesions involving the appendiceal orifice or ileocaecal valve.
* Patients with significant cardiorespiratory comorbidities which may limit their ability to undertake monitored anesthesia for the procedure.
* Poor performance status (Eastern Cooperation Oncology Group performance status ≥3).
* Pregnant women or those planning pregnancy or breastfeeding women.
* Uncorrectable coagulopathy defined by international normalized ratio (INR) > 1.5 or platelet count < 50000/µl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
En-bloc resection rate | 30 days
  Defined by complete macroscopic resection of the target neoplasia in one single specimen

SECONDARY OUTCOMES:
R0 resection rate | 30 days
  Defined by histologically margin negative resection (Both horizontal and vertical margins)
Curative resection rate | 30 days
  Defined by R0 resection and fulfilling existing histological curative resection criteria based on JGES guidelines
Adverse event rate | 30 days
  Overall adverse event rate, according to ASGE lexicon
Rate of adverse event - hemorrhage | 30 days
  Rate of intraprocedural and post procedural delayed hemorrhage
Rate of adverse event - perforation | 30 days
  Rate of intraprocedural and post procedural delayed perforation
Rate of adverse event - post-ESD coagulation syndrome | 30 days
  Defined by post-procedural abdominal pain and systemic inflammatory response

OTHER OUTCOMES:
Procedure time | 1 day
  Duration of ESD
Device dysfunction | 1 day
  Failure of device to continue the procedure
Need for change to other device | 1 day
  Rate of changing to other ESD knife

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided